CLINICAL TRIAL: NCT03074422
Title: Effectiveness and Reliability of Hypnosis in Stereotaxy
Acronym: ERST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marco Vincenzo Corniola, Chief Medical Officer, University Hospital, Geneva
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01843
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Parkinson Disease; Tremor, Essential; Dystonia, Primary
Keywords: Functional neurosurgery; Pain management; Hypnosis; Stereotaxy; Parkinson disease; Essential tremor; Dystonia; Invasive monitoring of epilepsy
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Dystonic Disorders; Agnosia; Dystonia | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Patients will be randomly attributed to either the "hypnosis" group or the control group, by a randomization process. The investigators plan to allocate patients in two groups; in the first group, patients will undergo hypnosis during the fixation of the stereotactic frame. In the second group (control group), the frame disposal will be performed following the actual standard of care, with a LA performed during the procedure.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypsnosis (Experimental): During the fixation of the stereotactic frame, a single hypnosis session is performed by a certified senior anesthesiologist. Blood pressure, heart rate and respiratory rate are continuously monitored by the mean of a regular scope. Pain perceived during and after the procedure is quantifies by the mean of the Visual Analogue Scale (VAS) questionnaire. An open, standardized question will be asked to participants concerning feelings and thoughts about the frame fixation. Answers will be audio recorded. A standardized perceived distress questionnaire (PDI-13) will be performed.
  Interventions: Procedure: Hypnosis
- Control (No Intervention): Local anesthesia after clear and complete information of the procedure given the day prior to the surgery. In order to determine the pain perceived during the procedure, a VAS questionnaire will be used, directly after the frame disposal. The rest of the procédure is similar to the hypnosis group.

INTERVENTIONS:
Procedure: Hypnosis — Hypnosis session performed by a board certified senior anesthesiologist during the frame fixation on the patient's head.
  Arms: Hypsnosis

SUMMARY:
In certain neurosurgical procedures, the use of a stereotaxic frame is required. It is then possible to set a precise target (depending of the type of the surgery) to be reached by the surgeon. The fixation of the stereotactic frame on the awake patient's head is done under local anesthesia by screwing the frame directly into the skull. This procedure is reported as "painful" to "extremely painful" by patients. The objective of this study is to determine whether the hypnosis is effective in decreasing the pain perceived by the patient during the disposal of the stereotactic frame.

DETAILED DESCRIPTION:
The role of hypnosis (no sedative drug administered) and hypnosedative procedures (hypnosis with the adjunct of a sedative drug) during surgical procedures has been largely discussed during the past 10 years, and those techniques are now widely practiced in the surgical field, for example during thyroidectomies. In neurosurgery specifically, the successful use of hypnosedation during awake neurosurgical procedures has been recently reported, with a positive feedback from the patients, together with good results regarding extent of resection, in the case of brain lesions located in eloquent areas.

Since 1990, many research groups identified the existence of hypnosis-related phenomena and their influence on the pain signal perception. These authors show that there is a modulation of the anterior cingulate area activity together with modified interconnectivity with other critical regions involved in nociception. In this context, the potential of hypnosis in pain modulation and, more extensively, patient management in surgical anesthetics was established.

In various neurosurgical procedures, the use of a stereotactic frame is required; by using coordinates (x, y and z), which are computed and reported on the frame before the intervention, it is possible to set a precise target (dependent on the type of surgery) to be reached by the surgeon. For instance, during a Deep Brain Stimulation (DBS) performed in a patient suffering from Parkinson's disease (PD), the electrodes are introduced into the brain, deep down to the sub-thalamic nuclei (STN), which are situated in a very little area located in the upper brainstem. The mounting of the stereotactic frame on the patient's head is performed under local anesthesia (LA), as the patient is awake during the mounting procedure and later on during the surgical intervention. This mounting is done by screwing the device directly into the patient's skull, through the skin. This moment is reported as "painful" to "extremely painful" by patients, and most of them confess to keep a very unpleasant memory of the event, even several years after the procedure and despite the fact that the surgery had a positive effect on their functional outcome.

As exposed above, there is still room for improvement in the management of pain and comfort of patients undergoing functional procedures in neurosurgery, especially during the placement of the stereotactic frame. To our opinion, hypnosis could represent a serious therapy against pain and anxiety generated by the frame fixation, especially those whom facial expressions and feelings might be altered by their pathology (i.e. Parkinson's disease). In fact, this technique has already been abundantly reported as an important adjuvant to the management of pain and comfort during surgeries such as thyroidectomies) and resection of brain tumors.

The main objective of this study is to determine whether hypnosis is effective in decreasing the pain perceived by the patient during the placement of the stereotactic frame on the patient's head.

The secondary aims of this study are: 1) to measure the stress perceived during the procedure by submitting the patient to validated scores and 2) to evaluate the incidence of Post-traumatic Stress Disorder (PTSD), according to the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a stereotactic procedure as listed previously
* Patients ≥ 18 y.o.

Exclusion Criteria:

* Patients < 18 y.o.
* Patients unable to take decisions by their own
* Patients undergoing deep brain stimulation for obsessive-compulsive disease treatment
* Patients refusing to participate to the study
* Pregnancy
* Invasive monitoring of epilepsy
* Psychiatric comorbidity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Effect on pain | 2 years
  To determine whether the hypnosis is effective in decreasing the pain perceived by the patient during the placement of the stereotactic frame on the patient's head.

SECONDARY OUTCOMES:
Effect on the stress perceived during the procedure | 2 years
  To measure the stress perceived during the procedure by submitting the patient to validated scores .
Effect on the incidence of post-traumatic stress disorder | 2 years
  To evaluate the incidence of Post-traumatic Stress Disorder (PTSD), according to the DSM-IV criteria

CONTACTS AND LOCATIONS:
Overall Officials: Marco Corniola, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang DD, Lau D, Rolston JD, Englot DJ, Sneed PK, McDermott MW. Pain experience using conventional versus angled anterior posts during stereotactic head frame placement for radiosurgery. J Clin Neurosci. 2014 Sep;21(9):1538-42. doi: 10.1016/j.jocn.2014.02.009. Epub 2014 May 6. PMID 24814855
- [Background] Rahman M, Murad GJ, Mocco J. Early history of the stereotactic apparatus in neurosurgery. Neurosurg Focus. 2009 Sep;27(3):E12. doi: 10.3171/2009.7.FOCUS09118. PMID 19722814
- [Background] Murata J, Sawamura Y, Kitagawa M, Saito H, Kikuchi S, Tashiro K. [Minimally invasive stereotactic functional surgery using an intravenous anesthetic propofol and applying Image Fusion and AtlasPlan]. No To Shinkei. 2001 May;53(5):457-62. Japanese. PMID 11424357
- [Background] Venkatraghavan L, Manninen P, Mak P, Lukitto K, Hodaie M, Lozano A. Anesthesia for functional neurosurgery: review of complications. J Neurosurg Anesthesiol. 2006 Jan;18(1):64-7. doi: 10.1097/01.ana.0000181285.71597.e8. PMID 16369142
- [Background] Stokes MA, Soriano SG, Tarbell NJ, Loeffler JS, Alexander E 3rd, Black PM, Rockoff MA. Anesthesia for stereotactic radiosurgery in children. J Neurosurg Anesthesiol. 1995 Apr;7(2):100-8. doi: 10.1097/00008506-199504000-00005. PMID 7772962
- [Background] Benabid AL, Chabardes S, Mitrofanis J, Pollak P. Deep brain stimulation of the subthalamic nucleus for the treatment of Parkinson's disease. Lancet Neurol. 2009 Jan;8(1):67-81. doi: 10.1016/S1474-4422(08)70291-6. PMID 19081516
- [Background] Benabid AL, Chabardes S, Seigneuret E, Fraix V, Krack P, Pollak P, Xia R, Wallace B, Sauter F. Surgical therapy for Parkinson's disease. J Neural Transm Suppl. 2006;(70):383-92. doi: 10.1007/978-3-211-45295-0_58. PMID 17017557
- [Background] Chevrier E, Fraix V, Krack P, Chabardes S, Benabid AL, Pollak P. Is there a role for physiotherapy during deep brain stimulation surgery in patients with Parkinson's disease? Eur J Neurol. 2006 May;13(5):496-8. doi: 10.1111/j.1468-1331.2006.01298.x. PMID 16722975
- [Background] Fraix V, Pollak P, Chabardes S, Ardouin C, Koudsie A, Benazzouz A, Krack P, Batir A, Le Bas JF, Benabid AL. [Deep brain stimulation]. Rev Neurol (Paris). 2004 May;160(5 Pt 1):511-21. doi: 10.1016/s0035-3787(04)70980-7. French. PMID 15269668
- [Background] Benabid AL, Pollak P, Hommel M, Gaio JM, de Rougemont J, Perret J. [Treatment of Parkinson tremor by chronic stimulation of the ventral intermediate nucleus of the thalamus]. Rev Neurol (Paris). 1989;145(4):320-3. French. PMID 2660224
- [Background] Cojan Y, Waber L, Schwartz S, Rossier L, Forster A, Vuilleumier P. The brain under self-control: modulation of inhibitory and monitoring cortical networks during hypnotic paralysis. Neuron. 2009 Jun 25;62(6):862-75. doi: 10.1016/j.neuron.2009.05.021. PMID 19555654
- [Background] Zemmoura I, Fournier E, El-Hage W, Jolly V, Destrieux C, Velut S. Hypnosis for Awake Surgery of Low-grade Gliomas: Description of the Method and Psychological Assessment. Neurosurgery. 2016 Jan;78(1):53-61. doi: 10.1227/NEU.0000000000000993. PMID 26313220
- [Background] Tykocki T, Kornakiewicz A, Mandat T, Nauman P. Pain perception in patients with Parkinson's disease. J Clin Neurosci. 2013 May;20(5):663-6. doi: 10.1016/j.jocn.2012.05.043. Epub 2013 Feb 26. PMID 23485408
- [Background] Watson R, Leslie K. Nerve blocks versus subcutaneous infiltration for stereotactic frame placement. Anesth Analg. 2001 Feb;92(2):424-7. doi: 10.1097/00000539-200102000-00028. PMID 11159245
- [Background] Bellinghausen L, Collange J, Botella M, Emery JL, Albert E. [Factorial validation of the French scale for perceived stress in the workplace]. Sante Publique. 2009 Jul-Aug;21(4):365-73. French. PMID 20101815
- [Background] Jehel L, Brunet A, Paterniti S, Guelfi JD. [Validation of the Peritraumatic Distress Inventory's French translation]. Can J Psychiatry. 2005 Jan;50(1):67-71. doi: 10.1177/070674370505000112. French. PMID 15754668
- [Derived] Catalano Chiuve S, Momjian S, Wolff A, Corniola MV. Effectiveness and reliability of hypnosis in stereotaxy: a randomized study. Acta Neurochir (Wien). 2024 Feb 27;166(1):112. doi: 10.1007/s00701-024-05943-0. PMID 38411747